CLINICAL TRIAL: NCT02776046
Title: Individualized Perioperative Open-luna Ventilatory Strategy With High Versus Conventional Inspiratory Oxygen Fraction (iPROVE-O2). A Comparative, Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Individualized Perioperative Open-lung Ventilatory Strategy With High Versus Conventional Inspiratory Oxygen Fraction (iPROVE-O2).
Acronym: iPROVE-O2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: Hospital La Fe de Valencia (Unknown); Hospital General Universitario de Valencia (Other); Hospital de Manises (Other); Hospital de Elche (Unknown); Hospital de Villajoyosa (Unknown); Hospital San Pau de Barcelona (Unknown); Hospital Clinic of Barcelona (Other); Hospital Germans Tríes i Pujol de Badalona (Unknown); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital Gregorio Marañon de Madrid (Unknown); Hospital Ramón y Cajal de Madrid (Unknown); Hospital Puerta de Hierro de Majalahonda (Unknown); Hospital Universitario Fundación Alcorcón (Other); Hospital Virgen del Rocío de Sevilla (Unknown); Hospital Son Espases de Mallorca (Unknown); Hospital Dr. Negrin de la Palmas (Unknown); Hospital Nuestra Señora de la Candelaria de Santa Cruz de Tenerife (Unknown); Hospital de Leon (Other Government); Hospital POVISA de Vigo (Unknown); Hospital Álvaro Cunqueiro de Vigo (Unknown); Hospital de Albacete (Unknown); Hospital Principe de Asturias de Madrid (Unknown); Hospital Miguel Servet de Zaragoza (Unknown); Hospital General de Ciudad Real (Other); Hospital Río Hortega de Valladolid (Unknown)
Responsible Party: Principal Investigator, Carlos Ferrando, MD,PhD, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: iPROVE-O2
Record Dates: First submitted 2016-05-15; First posted 2016-05-18 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Hyperoxia; Postoperative Complication; Surgical Site Infection
Keywords: Oxygen, surgical site infection, postoperative complication, recruitment maneuvers, open lung strategy
MeSH Terms: conditions — Hyperoxia; Postoperative Complications; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High FiO2 (Experimental): Intraoperatively ventilated patients with a tidal volume (VT) of 8 ml / kg of ideal body weight, and a FiO2 of 0.8. After intubation, all patients were conduct an alveolar recruitment maneuver (MRA) and PEEP level individualized spanned (see Calculation of optimal PEEP). Every 40 minutes will be assessed the need to adjust the level of PEEP by evaluating the dynamic compliance of the respiratory system (Crs). Faced with a decline in Crs> 10% a new MRA and optimal PEEP setting will be assessed.
  Postoperatively 3h with 0.8 FiO2 and individualized CPAP
  Interventions: Drug: High FiO2
- Conventional FiO2 (Active Comparator): Intraoperatively ventilated patients with a tidal volume (VT) of 8 ml / kg of ideal body weight, and a FiO2 of 0.3. After intubation, all patients were conduct an alveolar recruitment maneuver (MRA) and PEEP level individualized spanned (see Calculation of optimal PEEP). Every 40 minutes will be assessed the need to adjust the level of PEEP by evaluating the dynamic compliance of the respiratory system (Crs). Faced with a decline in Crs> 10% a new MRA and optimal PEEP setting will be assessed.
  Postoperatively 3h with 0.3 FiO2 and individualized CPAP
  Interventions: Drug: Conventional FiO2

INTERVENTIONS:
Drug: High FiO2 — High FiO2 with a perioperative open lung strategy
  Arms: High FiO2
Drug: Conventional FiO2 — Conventional FiO2 with a perioperative open lung strategy
  Arms: Conventional FiO2

SUMMARY:
The iPROVE-O2 trial aims at comparing the efficacy of high and conventional FiO2 within a perioperative individualized ventilatory strategy to reduce the overall incidence of SSI.

ELIGIBILITY:
Inclusion Criteria:

* Age not less than 18
* Planned abdominal surgery> 2 hours.
* Signed informed consent for participation in the study.

Exclusion Criteria:

* Age less than 18 years.
* Pregnant or breast-feeding.
* Patients with BMI >35.
* Syndrome of moderate or severe respiratory distress: PaO2/FiO2 < 200 mmHg.
* Heart failure: NYHA IV.
* Hemodynamic failure: CI <2.5 L/min/m2 and / or requirements before surgery ionotropic support.
* Diagnosis or suspicion of intracranial hypertension (intracranial pressure> 15 mmHg).
* Mechanical ventilation in the last 15 days.
* Presence of pneumothorax. Presence of giant bullae on chest radiography or computed tomography (CT).
* Patient with preoperatively CPAP.
* Participation in another experimental protocol at the time of intervention selection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | seven postoperative days

SECONDARY OUTCOMES:
Systemic complications | seven postoperative days
Pulmonary complications | seven postoperative days
Systemic and pulmonary complications | thirty postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Javier Belda, Md, PhD, Study Director — Department of Anesthesia and Critical Care; Hospital Clinico Universitario
Locations (1):
- Department of Anesthesia and Critical Care; Hospital Clinico Universitario, Valencia, Spain

REFERENCES:
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Background] Belda FJ, Aguilera L, Garcia de la Asuncion J, Alberti J, Vicente R, Ferrandiz L, Rodriguez R, Company R, Sessler DI, Aguilar G, Botello SG, Orti R; Spanish Reduccion de la Tasa de Infeccion Quirurgica Group. Supplemental perioperative oxygen and the risk of surgical wound infection: a randomized controlled trial. JAMA. 2005 Oct 26;294(16):2035-42. doi: 10.1001/jama.294.16.2035. PMID 16249417
- [Background] Meyhoff CS, Wetterslev J, Jorgensen LN, Henneberg SW, Hogdall C, Lundvall L, Svendsen PE, Mollerup H, Lunn TH, Simonsen I, Martinsen KR, Pulawska T, Bundgaard L, Bugge L, Hansen EG, Riber C, Gocht-Jensen P, Walker LR, Bendtsen A, Johansson G, Skovgaard N, Helto K, Poukinski A, Korshin A, Walli A, Bulut M, Carlsson PS, Rodt SA, Lundbech LB, Rask H, Buch N, Perdawid SK, Reza J, Jensen KV, Carlsen CG, Jensen FS, Rasmussen LS; PROXI Trial Group. Effect of high perioperative oxygen fraction on surgical site infection and pulmonary complications after abdominal surgery: the PROXI randomized clinical trial. JAMA. 2009 Oct 14;302(14):1543-50. doi: 10.1001/jama.2009.1452. PMID 19826023
- [Background] Greif R, Akca O, Horn EP, Kurz A, Sessler DI; Outcomes Research Group. Supplemental perioperative oxygen to reduce the incidence of surgical-wound infection. N Engl J Med. 2000 Jan 20;342(3):161-7. doi: 10.1056/NEJM200001203420303. PMID 10639541
- [Derived] Ferrando C, Librero J, Tusman G, Serpa-Neto A, Villar J, Belda FJ, Costa E, Amato MBP, Suarez-Sipmann F; iPROVE Network Group. Intraoperative open lung condition and postoperative pulmonary complications. A secondary analysis of iPROVE and iPROVE-O2 trials. Acta Anaesthesiol Scand. 2022 Jan;66(1):30-39. doi: 10.1111/aas.13979. Epub 2021 Sep 22. PMID 34460936
- [Derived] Ferrando C, Aldecoa C, Unzueta C, Belda FJ, Librero J, Tusman G, Suarez-Sipmann F, Peiro S, Pozo N, Brunelli A, Garutti I, Gallego C, Rodriguez A, Garcia JI, Diaz-Cambronero O, Balust J, Redondo FJ, de la Matta M, Gallego-Ligorit L, Hernandez J, Martinez P, Perez A, Leal S, Alday E, Monedero P, Gonzalez R, Mazzirani G, Aguilar G, Lopez-Baamonde M, Felipe M, Mugarra A, Torrente J, Valencia L, Varon V, Sanchez S, Rodriguez B, Martin A, India I, Azparren G, Molina R, Villar J, Soro M; iPROVE-O2 Network. Effects of oxygen on post-surgical infections during an individualised perioperative open-lung ventilatory strategy: a randomised controlled trial. Br J Anaesth. 2020 Jan;124(1):110-120. doi: 10.1016/j.bja.2019.10.009. Epub 2019 Nov 22. PMID 31767144
- [Derived] Ferrando C, Soro M, Unzueta C, Canet J, Tusman G, Suarez-Sipmann F, Librero J, Peiro S, Pozo N, Delgado C, Ibanez M, Aldecoa C, Garutti I, Pestana D, Rodriguez A, Garcia Del Valle S, Diaz-Cambronero O, Balust J, Redondo FJ, De La Matta M, Gallego L, Granell M, Martinez P, Perez A, Leal S, Alday K, Garcia P, Monedero P, Gonzalez R, Mazzinari G, Aguilar G, Villar J, Belda FJ; iPROVE-O2 Network Group. Rationale and study design for an individualised perioperative open-lung ventilatory strategy with a high versus conventional inspiratory oxygen fraction (iPROVE-O2) and its effects on surgical site infection: study protocol for a randomised controlled trial. BMJ Open. 2017 Jul 31;7(7):e016765. doi: 10.1136/bmjopen-2017-016765. PMID 28760799